CLINICAL TRIAL: NCT02181361
Title: The Efficacy and Safety of Hirudin Plus Aspirin Versus Warfarin in the Secondary Prevention of Cardioembolic Stroke Due to Nonvalvular Atrial Fibrillation: a Prospective Cohort Study
Brief Title: Hirudin Plus Aspirin in the Secondary Prevention of Cardioembolic Stroke Due to Nonvalvular Atrial Fibrillation
Status: Completed | Type: Observational
Sponsor: Xijing Hospital (Other)
Collaborators: Xi'an Central Hospital (Other); Shaanxi people's Hospital (Unknown); The Third Hospital of PLA (Unknown); Hanzhong Central Hospital (Other); Xianyang 215 hospital (Unknown); Yulin Second Hospital (Unknown); Yan'an University Affiliated Hospital (Other); Baoji Central Hospital (Other); Ankang Central Hospital (Other); Baoji People's Hospital (Unknown); Yan'an people's Hospital (Unknown); 451 Hospital (Unknown); Shangluo Central Hospital (Other); Central Hospital of China Railway 20th Bureau (Unknown); Xiangyang Central Hospital (Other); Xi'an Ninth Hospital (Unknown); Shangluo Second People's Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: Xijing-4-3
Record Dates: First submitted 2014-06-03; First posted 2014-07-03 (Estimated); Last update posted 2020-04-21 (Actual); Status verified 2013-09

CONDITIONS: Cardioembolic Stroke; Atrial Fibrillation
Keywords: atrial fibrillation; cardioembolic stroke; Hirudin; aspirin; warfarin
MeSH Terms: conditions — Embolic Stroke; Atrial Fibrillation | interventions — Hirudins; Aspirin; Warfarin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- hirudin plus aspirin: 14 days after stroke onset, patients in the hirudin plus aspirin group received natural hirudin 0.75g, three times a day and aspirin 100mg, once daily.
  Interventions: Drug: hirudin plus aspirin
- Warfarin: 14 days after stroke onset, patients in warfarin group were given an initial dose of 1.25mg of warfarin,once daily. 3 days later, INR of patients was checked every three days and the dose of warfarin was adjusted until reach the target range of 2 to 3. Since then INR monitoring was performed at 1, 2, 3, 6, 9, 12 months after stroke onset, targeting an INR between 2 and 3 and the dose of warfarin was adjusted accordingly.
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: hirudin plus aspirin — natural hirudin 0.75g, three times a day (Brand name: Maixuekang capsule, Guizhou Xinbang Pharmaceutical Co., China) and aspirin 100mg, once daily
  Groups: hirudin plus aspirin
Drug: Warfarin — an initial dose of 1.25mg once daily. Three days later, INR of patients was checked every three days and the dose of warfarin was adjusted until reach the target range of 2 to 3. Since then INR monitoring was performed at 1, 2, 3, 6, 9, 12 months after stroke onset, targeting an INR between 2 and 3 and the dose of warfarin was adjusted accordingly.
  Groups: Warfarin

SUMMARY:
To investigate the efficacy and safety of hirudin plus aspirin therapy compared with warfarin in the secondary prevention of cardioembolic stroke due to nonvalvular atrial fibrillation.

DETAILED DESCRIPTION:
For the patients with cardioembolic stroke due to atrial fibrillation,guidelines recommended warfarin as the secondary prevention therapy. But warfarin has its disadvantages such as risk of bleeding and the requirement of frequent INR monitoring. The underuse of warfarin is a prominent problem in China. In our study, patients with cardioembolic stroke were treated with hirudin plus aspirin or warfarin. The aim of our study was to compare efficacy and safety of hirudin plus aspirin and warfarin in secondary prevention of cardioembolic stroke due to nonvalvular atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

1. age of 18 or older with NVAF-related cardioembolic stroke
2. diagnosis of cardioembolic stroke conformed to the TOAST (Trial of Org 10172 in Acute Stroke Treatment) classification system in terms of the typical clinical presentation, neuroimaging profile, and vascular and cardiac evaluation
3. patients who were after 14 days of stroke onset and with stable clinical status.

Exclusion Criteria:

1. patients with rheumatic heart disease or history of heart valve surgery;
2. patients with acute coronary syndrome or percutaneous coronary intervention within 30 days previous to enrollment;
3. patients with active infective endocarditis;
4. patients with purpura disease or blood coagulation disorder;
5. patients who had active bleeding or the tendency to bleed;
6. patients with history of intracranial hemorrhage (ICH) or other serious bleeding events;
7. patients diagnosed with peptic ulcer disease within 30 days previous to enrollment;
8. patients who had esophageal varices;
9. patients who had trauma or major surgery within 30 days previous to enrollment or patients who planned to have major surgery;
10. patients with persistent blood pressure of 180/100mmHg or greater with or without anti-hypertension treatment;
11. patients who need chronic anticoagulant treatment due to disorders other than AF;
12. patients with severe liver and kidney dysfunction;
13. patients who were allergic to warfarin, aspirin or hirudin;
14. female patients who are pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cardioembolic stroke patients due to nonvalvular atrialf ibrillation.
Sampling Method: Probability Sample
Enrollment: 239 (Actual)
Dates: Start 2014-06; Primary Completion 2016-12 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Efficacy outcome event: the recurrence of cardioembolic stroke | One year after stroke onset
  To compare the recurrence of cardioembolic stroke in hirudin plus aspirin group and the warfarin group.

OTHER OUTCOMES:
Safety outcome events | One year after stroke onset
  Intracranial hemorrhage and other bleeding events, any death and other serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: wen jiang, MD,PhD, Study Chair — The Department of Neurology , Xijing Hospital
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China